CLINICAL TRIAL: NCT05236465
Title: A 3-day Course for Adults With Chronic Fatigue Syndrome/Myalgic Encephalopathy (CFS/ME): a Randomized Controlled Trial
Brief Title: A 3-day Course for CFS/ME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: University of Oslo (Other); Haukeland University Hospital (Other); Lørenskog municipality (Unknown); The Research Council of Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 394844
Record Dates: First submitted 2022-02-04; First posted 2022-02-11 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Chronic Fatigue Syndrome; Myalgic Encephalomyelitis
Keywords: Health education; Chronic Fatigue Syndrome/Myalgic Encephalopathy (CFS/ME); RCT; 3-day Course; Physical function; Fatigue; Cognitive techniques; Behavioral activation
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Health Education; Fatigue | interventions — Waiting Lists

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial, in which participants are randomly allocated to either the intervention group or to the waiting list control group.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The intervention group vs. waiting list control group status will be known to the participants and the personnel delivering the 3-day course. However, the investigator and outcome assessor will be masked to the conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A 3-day course (Experimental): The course consists of teaching in basic psychology, stress physiology and practice of a specific technique with self-instructions and visualization in a group setting by non-health personnel
  Interventions: Behavioral: A 3-day course
- Waiting list (Active Comparator): Treatment as usual (TAU)
  Interventions: Behavioral: Waiting list

INTERVENTIONS:
Behavioral: A 3-day course — The course is built on the LP manual (Parker, 2013) and includes stress theory, Positive Psychology and knowledge about regulating thoughts, feelings and behavior, and through that positively influencing physiology.
  Arms: A 3-day course
Behavioral: Waiting list — Treatment as usual (TAU) in the first 10 weeks. After 10 weeks: Behavioural: A 3-day course. The course is built on the LP manual (Parker, 2013) and includes stress theory, Positive Psychology and knowledge about regulating thoughts, feelings and behavior, and through that positively influencing physiology.
  Arms: Waiting list

SUMMARY:
Chronic fatigue syndrome/Myalgic encephalomyelitis (CFS/ME) can be a serious and disabling condition with a heavy symptom burden and low function. Work disability is common, and social life dramatically affected. CFS/ME is a challenging health problem as well as a societal problem.

In recent years, a doubling of the number of patients with a CFS/ME diagnoses has been reported in Norway. The patient group represents a challenge for the health care system, the municipality, and the Norwegian Labour and Welfare Organization (NAV). According to new figures, the NAV pays 100 million Norwegian Kroner (NOK) each month in permanently incapacitated expenses for people with CFS/ME. Municipalities have expenses in form of care, rehabilitation and other measures.

There is a lack of effective treatment for CFS/ME. Evidence-based knowledge is highly needed.

If the 3-day course shows promising effects, this could have positive consequences for patients, relatives and health personnel, but also financially for the society and the municipality.

DETAILED DESCRIPTION:
This is a randomized controlled trial (RCT) to investigate potential effects (positive and negative) of a 3-day course with follow-up for 100 adults with CFS/ME.

The 3-day course used in this trial is named the Lightning Process (LP). The course is built on the LP manual (Parker, 2013) and includes stress theory, Positive Psychology and knowledge about regulating thoughts, feelings and behavior, and through that positively influencing physiology.

Positive and negative effects of the course on symptoms, disability and quality of life will be investigated, and a long-term follow-up of work participation conducted.

Any adverse events experienced during or after the 3-day course will be handled according to protocol.

ELIGIBILITY:
Inclusion Criteria:

* CFS/ME diagnosis based on the Canada Consensus Criteria.
* At least 50% out of school/work.
* Readiness to change (corresponding to the preparation phase in transtheoretical model)
* Has given informed consent.

Exclusion Criteria:

* Assessed by a General Practitioner (GP):
* Underlying physical illness or mental disorder that may explain the symptoms.
* Suicide risk/previous suicide attempts.
* Pregnancy.
* Bedridden and in need of continuous care.
* Insufficient Norwegian speaking or writing skills to participate in the 3-day course and fill out questionnaires.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Physical function | 10 weeks after the 3-day course
  Measured through the Short Form Health Survey (SF-36), physical function, a scale that measures physical function with questions relating to ability to perform physical activity. The instrument contains 10 items with three options on each question. The score range is 0 -100, where 100 is equivalent to no disability.

SECONDARY OUTCOMES:
Fatigue | 6 months after the 3-day course
  Measured through the Chalder Fatigue Questionnaire, an instrument that measures fatigue severity, both on mental and physical fatigue in the last month. The instrument contains 11 items with four different response options in each question. The scale ranges from 0-33, where higher score indicates greater fatigue.
Pain on a daily basis | 6 months after the 3-day course
  Measured through the Brief Pain Inventory, an instrument measuring pain and its allied aspects. The instrument contains 11 items with numeric rating from 0-10, where higher score indicates more severe pain.
Post-Exertional Malaise | 6 months after the 3-day course
  Measured through A Brief Questionnaire to Assess Post-Exertional Malaise, an instrument that measures symptoms after activity. The instrument contains 10 items, with options ranging from 0-4, where a higher score indicates more severity.
Mental wellbeing | 6 months after the 3-day course
  Measured trough the Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS), an instrument that measures mental wellbeing. The instrument contains 14 items, with 5 response categories, summed to provide a single score. Higher score indicates better wellbeing.
Overall improvement | 6 months after the 3-day course
  Measured through the Patient Global Impression of Change (PGIC) with one single item that measures change in function, symptoms and quality of life. The instrument has seven possible options ranging from very much better to very much worse.
Sick leave | 24 months after the 3-day course
  Register data from the Norwegian Labour and Welfare Administration (NAV) on sick leave, benefits, diagnoses from 12 months before the 3-day course and 24 months after the 3-day course.

CONTACTS AND LOCATIONS:
Overall Officials: Leif Edward Ottesen Kennair, PhD prof, Principal Investigator — NTNU, Department of Psychology
Locations (1):
- Department of Psychology, NTNU, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, along with the intervention protocol, will be published and publicly available. Registry data will not be shared as this is not allowed to share according to Norwegian law. However, Anonymized data can be shared with other researchers on reasonable request for use in specific research projects on CFS/ME after this study has been published. Due to privacy concerns, the complete data files will not be shared online.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The study protocol and the intervention protocol will be publicly available upon study completion.
Access Criteria: Anonymized data involving self-report data will be shared upon reasonable request from other researchers for use in specific research projects on CFS/ME when the main analyses are completed and published.